CLINICAL TRIAL: NCT05125367
Title: Ten-Year Outcomes of Randomized Comparison of Coronary Artery Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease: The BEST Extended 10 Y Follow-up
Brief Title: Ten-Year Outcomes of Randomized Comparison of Coronary Artery Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease
Acronym: BEST Extended
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV 2021-03
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: multivessel coronary artery disease; percutaneous coronary intervention; coronary artery bypass graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multivessel coronary artery disease: From BEST trial study population_NCT00997828
  Interventions: Procedure: coronary stent implantation; Procedure: bypass grafting

INTERVENTIONS:
Procedure: coronary stent implantation — coronary stent implantation using everolimus-eluting balloon expandable stents
Procedure: bypass grafting — coronary artery bypass graft

SUMMARY:
The primary objective of the BEST extended 10Y follow-up study is to compare the safety and effectiveness of coronary stent implantation using everolimus-eluting balloon-expandable stents with bypass grafting for the treatment of multivessel coronary artery disease at minimum of 10 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Angiographically confirmed multivessel coronary artery disease [critical (>70%) lesions in at least two major epicardial vessels (≥ 2.0mm in diameter) at least two separate coronary artery territories (the right coronary artery (RCA), left circumflex artery (LCX) and left anterior descending (LAD)] and are expected to be equally treatable with PCI(Percutaneous Coronary Intervention) or CABG(coronary artery bypass graft) by interventionalists and surgeons at the investigating site.
3. Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia
4. Geographically accessible and willing to come in for required study visits
5. Signed informed consent.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications:

   * Heparin
   * Aspirin
   * Both Clopidogrel and TIclopidine
   * Sirolimus, paclitaxel, ABT 578
   * Stainless steel and/or
   * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
2. Severe congestive heart failure (class III or IV according to New York Heart Association (NYHA) Functional Classification, or pulmonary edema) at the time of enrollment. The degree of left ventricular ejection fraction is not considered as an index of exclusion.
3. Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stent).
4. Prior CABG surgery
5. Prior PCI with DES implantation within 1 year
6. Two or more chronic total occlusions in major coronary territories
7. Acute ST-elevation myocardial infarction(Q-wave) within 72 hours prior to enrollment requiring revascularization.
8. Abnormal creatine kinase (CK > 2x normal) and/or abnormal CK-MB levels and/or elevated Troponin levels at time of randomization. When the cardiac enzyme is returned to normal, those can be enrolled.
9. Previous stroke within 6 months or patients with stroke at more than 6 months with significant residual neurologic involvement.
10. Extra-cardiac illness that is expected to limit survival to less than 2 years; e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease.
11. Prior history of significant bleeding (within the previous 6 months) that might be expected to occur during CABG or PCI/DES(drug eluting stent) related anticoagulation.
12. Contraindication either CABG or PCI/DES because of a coexisting clinical condition
13. Intolerance or contraindication to aspirin or both clopidogrel and ticlopidine
14. Suspected pregnancy.
15. Concurrent enrollment in another clinical trial
16. Left main stenosis (at least 50% diameter stenosis)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The BEST trial study population: patients with multivessel coronary artery disease treated by coronary stent implantation using everolimus-eluting balloon expandable stents or the bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) including all-cause mortality, myocardial infarction, or target vessel revascularization (TVR) | 10-year
  A composite endpoint(MACE) is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.
  Definitions for primary and secondary clinical outcomes are consistent with those used in the original BEST trial protocol(NCT00997828).

SECONDARY OUTCOMES:
Composite of death, myocardial infarction, or stroke | 10-year
Composite of death, myocardial infarction, stroke, or any repeat revascularization | 10-year
All-cause death | 10-year
Myocardial infarction | 10-year
Stroke | 10-year
Target vessel revascularization (TVR) | 10-year
Any repeat revascularization | 10-year

CONTACTS AND LOCATIONS:
Locations (24):
- China (2):
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhongshan Hospital, Shanghai
- Sarawak General Hospital, Kuching, Malaysia
- South Korea (20):
  - Asan Medical Center, Seoul, Songpa-gu
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Inje University Pusan Paik Hospital, Pusan
  - Gangnam Severance Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee J, Ahn JM, Kim H, Choi Y, Jo S, Kang DY, Kim MJ, Hur SH, Park HJ, Tresukosol D, Kang WC, Kwon HM, Rha SW, Lim DS, Jeong MH, Lee BK, Huang H, Lim YH, Bae JH, Kim BO, Ong TK, Ahn SG, Chung CH, Park DW, Park SJ; BEST Extended Follow-up Study investigators. Long-term outcomes of intravascular ultrasound-guided percutaneous coronary intervention versus coronary artery bypass grafting for multivessel coronary artery disease. Heart. 2025 Sep 11;111(19):918-924. doi: 10.1136/heartjnl-2024-325107. PMID 40368452
- [Derived] Ahn JM, Kang DY, Yun SC, Ho Hur S, Park HJ, Tresukosol D, Chol Kang W, Moon Kwon H, Rha SW, Lim DS, Jeong MH, Lee BK, Huang H, Hyo Lim Y, Ho Bae J, Ok Kim B, Kiam Ong T, Gyun Ahn S, Chung CH, Park DW, Park SJ; BEST Extended Follow-Up Study Investigators. Everolimus-Eluting Stents or Bypass Surgery for Multivessel Coronary Artery Disease: Extended Follow-Up Outcomes of Multicenter Randomized Controlled BEST Trial. Circulation. 2022 Nov 22;146(21):1581-1590. doi: 10.1161/CIRCULATIONAHA.122.062188. Epub 2022 Sep 19. PMID 36121700